CLINICAL TRIAL: NCT03970369
Title: Motivated to Move: A Randomized Pilot Study to Determine the Feasibility of Self-Monitoring on Self-Perceptions Towards Physical Activity in Youth
Brief Title: Motivated to Move: A Study to Determine the Feasibility of Self-Monitoring Physical Activity in Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: M2M-5234
Record Dates: First submitted 2019-05-16; First posted 2019-05-31 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Chronic Disease; Child; Adolescent
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monitor (Experimental): Activity monitoring with feedback. Participants in the Monitor group will wear a step counter to track if the activity prescription is being met.
  Interventions: Behavioral: Usual care; Behavioral: Monitor
- Usual care (Active Comparator): All children will receive the usual care, which includes personalized goals and an activity prescription. Participants in the usual care group will not receive a step counter.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Usual care — Personalized goals and an activity prescription.
Behavioral: Monitor — Participants wear a step counter to track activity goals.
  Arms: Monitor

SUMMARY:
Children with a medical condition don't get enough exercise, which can lead to even more health problems in childhood and adulthood. To help patients be more active, the McMaster Children's Hospital has an Exercise Medicine Clinic, where kids with any medical condition can get help from doctors and exercise specialists to safely become more active. The Exercise Medicine Clinic works with kids that have arthritis, inflammatory bowel disease, cystic fibrosis, cerebral palsy, cancer, diabetes, and a lot of other conditions. So far, most of the kids that go to the Exercise Medicine Clinic show improved fitness levels, but other kids don't seem to improve at all. These differences in improvements probably relate to how much physical activity the patients do on a regular basis. What is not known is exactly how to motivate the patients to be more active. In the Motivated to Move study, the investigators are going to learn more about how technology can be used to help kids feel more motivated to be active. The purpose of the Motivated to Move study is to see if it's feasible for patients to use step trackers over a 6-month period as part of the care patients receive at the Exercise Medicine Clinic. The results from the study will be used to see how the step tracking worked and to design a larger study that compares motivation to be physically active between children who wear and don't wear step trackers.

DETAILED DESCRIPTION:
The Motivated to Move study is a single-centre, pilot randomized controlled trial that has been designed based on experience to be minimally intrusive to the busy lives of patients and families. As part of a typical Exercise Medicine Clinic (EXMED) visit, children receive an individualized physical activity prescription to follow for the next three months. Participants of Motivated to Move will receive this prescription and be randomized to either a MONITOR group or USUAL CARE. The monitor group will wear a step counter to track if participants are meeting the activity prescription. This study will determine if this step counter affects the participants' motivation, self regulation, and perceived competence with respect to physical activity, which will be measured with questionnaires.

Participants enrolled in the Motivated to Move study will undergo a total of 3 study visits over the course of 6 months. All study visits will take place as part of the patient's EXMED clinic visits, which are scheduled every 3 months. Eligible patients will be identified by a member of the EXMED team and be invited to learn more about the Motivated to Move study. All interested patients will have the opportunity to speak with the study research coordinator about the study. Consent and/or assent (as appropriate) will be obtained from patients who would like to participate in the Motivated to Move study. Upon providing consent, all participants will undergo a similar protocol, which includes a total of 3 study visits that coincide with a clinic appointment:

At the baseline study visit all participants will be asked to complete a series of questionnaires related to motivation, self-regulation, and perceived competence with respect to physical activity. Participants will then meet with the Exercise Physiologist to perform a fitness assessment. Next, participants will discuss the results of the fitness assessment and develop goals with the Kinesiologist. Participants will also receive a detailed, individualized physical activity prescription for the next three months. At the end of the clinic visit, the research assistant will randomize each participant into one of two groups: no activity monitoring (USUAL CARE) or activity monitoring with feedback (MONITOR). All participants, regardless of group, will be given an accelerometer (research-grade physical activity monitor), which is worn around the waist for 7 days. This protocol (with the exception of randomization) will be repeated at the participant's 3-month and 6-month study visits. Upon completion of the 3 study visits, participants will complete a brief questionnaire to assess the acceptability of the activity monitoring and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Newly referred patients to the Exercise Medicine Clinic (i.e. either first or second visit)
* 8-17 years old

Exclusion Criteria:

* Inability to communicate in English

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2019-06-20 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Estimate the recruitment rates | 10 months
  The recruitment rate will be determined by calculating the proportion of eligible children who enroll in the study over the estimated 10-month recruitment period
Investigate retention to the trial at the 3-month follow up visit | 3 months
  Proportion of participants who remained enrolled in the study (regardless of data completeness) at 3-months
Investigate retention to the trial at 6-month follow up visit. | 6 months
  Proportion of participants who remained enrolled in the study (regardless of data completeness) at 6-months.
Determine the feasibility of activity monitoring over the first 3 months | 3 months
  The participants' compliance wearing the activity monitor will be measured by determining the % of days participants wore the monitor over the first 3 months
Determine the feasibility of activity monitoring over 6 months | 6 months
  The participants' compliance wearing the activity monitor will be measured by determining the % of days participants wore the monitor over 6 months
Determine the acceptability of activity monitoring | 6 months
  A brief survey will be used at the final visit (6-mo) to assess the acceptability of activity monitoring

SECONDARY OUTCOMES:
Change in self-regulation and motivation | baseline, 3- and 6-months
  Measured using Behavioural Regulation in Exercise Questionnaire 3 (BREQ-3). The BREQ-3 includes 4 items (responses 0-4) for each of the following 6 dimensions: amotivation, external regulation, introjected regulation, identified regulation, integrated regulation, intrinsic regulation. Dimensions are calculated by the average score on the 4 corresponding items.
Change in perceived competence in physical activity | baseline, 3- and 6-months
  Measured using the Self-Perceived Competence in Physical Education Scale. Responses (1-7) of 4 items will be averaged. A higher score indicates greater perceived competence.
Change in autonomy (supportive vs. controlling) | baseline, 3- and 6-months
  Patients' perceptions of the degree to which their health care providers are autonomy supportive vs. controlling. Measured using the Health Care Climate questionnaire. Responses (1-7) on 6 items are averaged. A higher score indicates higher perception of supportive autonomy.
Change in physical activity | Baseline, 3- and 6-months
  1-week free-living physical activity measured via accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Obeid, PhD, Principal Investigator — McMaster University
Locations (1):
- Exercise Medicine Clinic at McMaster Children's Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No